CLINICAL TRIAL: NCT04482465
Title: Omega 3 and Vitamin D Dosage in a Population With Moderate to High Risk of Age-related Macular Degeneration
Brief Title: Omega 3 and Vitamin D Dosage in a Population With Moderate to High Risk of AMD
Acronym: OVID-AMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UZLeuven S59711
Record Dates: First submitted 2020-07-07; First posted 2020-07-22 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2020-07

CONDITIONS: Age-related Macular Degeneration; Vitamin D Deficiency
Keywords: micronutrients
MeSH Terms: conditions — Macular Degeneration; Vitamin D Deficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: epidemiological intervention pilot study
Masking Description: blood results were communicated to each participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pilot study 1 arm (Other): 50 subjects with no AMD or early AMD, aged over 55, at moderate-to-high risk for AMD based on a simplified AMD risk assessment scale score > or = 10, not taking vitamin D or trace nutriënt containing supplements
  Interventions: Diagnostic Test: blood sample

INTERVENTIONS:
Diagnostic Test: blood sample — blood sample to determine omega6/omega 3 ratio, EPA, DHA, zinc, cupric oxide, vitamine D

SUMMARY:
Objectives: The investigators conducted a prospective study in Belgium with the objective to determine the proportion of subjects identified at moderate-to-high risk for AMD, based on the STARS® questionnaire, in need of nutritional supplementation by assessing their vitamin D, zinc oxide and fatty acid profile status.

Methods: This multicentre epidemiological intervention pilot study involved 50 Belgian subjects with no AMD or early AMD, aged over 55, at moderate-to-high risk for AMD based on a simplified AMD risk assessment scale (STARS®) score ≥ 10, not taking vitamin D or trace nutrient containing supplements. Outcome data was collected during a one-time subject interview comprising of clinical eye examinations (typically visual acuity), the STARS® questionnaire, visual acuity assessment, an OCT scan on the macula, and fundus photography. Blood samples were collected from the patients and serum analysis was performed to determine the levels of omega-6 to omega-3 ratio, EPA and DHA, zinc and cupric oxide, and vitamin D, recognised as key nutrients involved in AMD pathophysiology.

DETAILED DESCRIPTION:
Study population This pilot study is a multicentre epidemiological intervention study of exploratory nature, hence no power calculation was performed, aiming to demonstrate trends. The study includes 50 subjects without a control group.

The inclusion criteria of the 50 subjects are: people over 55 years old, with a STARS® score ≥10 (moderate-to-high risk for AMD). Individuals with a STARS® score <10, or taking nutritional supplements containing vitamin D or trace nutrients in the 4 months prior to enrolment, and people with grade-3 or grade-4 AMD scores according to the AREDS simplified scale, were excluded from the study.

Study Design and Procedures The study was conducted in accordance to the GCP and Declaration of Helsinki principles, and the study protocol and all relevant study documents were submitted for review to the UZ Leuven Ethics Committee. Informed consent form was obtained from the subjects prior to their enrolment in the study. All information collected was kept confidential and anonymized and used exclusively for the purposes of this study in compliance with the applicable personal data protection and processing laws.

The study was completed within a single visit. Outcome data was collected during a one-time subject interview comprising of clinical eye examinations (typically visual acuity), the STARS® questionnaire, visual acuity assessment, an OCT scan on the macula, and fundus photography. Blood samples were collected using a Vacutainer system with 1 purple EDTA tube and 2 red tubes to assay for omega-3 fatty acids, EPA and DHA as well as omega-6 for the calculation of the omega-6:omega-3 (Ω6:Ω3) ratio, vitamin 25(OH)D, zinc oxide and cupric oxide. Samples were analysed by the RP Lab, Rue Emile Francqui 7, 1435 Mont-Saint-Guibert, Belgium (www.rplab.be).

Data Analysis The data were tested for normality using the Chi-Squared Goodness-of-Fit test. Data distribution was not normal for some of the assayed micronutrients, thus all data were analysed to identify trends using subject proportions (%) and descriptive statistics for not normally distributed data: median ± MAD (median absolute deviation).

ELIGIBILITY:
Inclusion Criteria:

* age over 55
* STARS score > or = 10 (moderate to high risk for AMD)

Exclusion Criteria:

* STARS score < 10
* persons taking nutritional supplements containing vitamin D or trace nutrients in the 4 months prior to enrollment
* persons with grade-3 or grade-4 AMD scores according to the AREDS simplified scale

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
concentration of vitamin D | at the time of the procedure
  vitamin D deficiency

SECONDARY OUTCOMES:
concentration of fatty acids | at the time of the procedure
  omega 6/omega 3 ratio, DHA, EPA
concentration of zinc oxide | at the time of the procedure
  in µg/L

CONTACTS AND LOCATIONS:
Overall Officials: Julie Jacob, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No
results will be published

REFERENCES:
- [Derived] Jacob J, Mangelschots E, Michez M, Sanak SN, Leys A. Cross-Sectional Study on Vitamin D, Zinc Oxide and Fatty Acid Status in a Population with a Moderate to High Risk of AMD Identified by the STARS(R) Questionnaire. Ophthalmol Ther. 2021 Jun;10(2):299-311. doi: 10.1007/s40123-021-00335-4. Epub 2021 Feb 23. PMID 33620690

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT04482465/Prot_SAP_000.pdf